CLINICAL TRIAL: NCT03654339
Title: Comparison of Conventional vs Microsurgical Method for Root Coverage by Lateral Displacement Flap
Brief Title: Microsurgical vs Macro Surgical Approach for Grade II Gingival Recessions Employing Laterally Repositioned Flap
Acronym: CCMMRCLDF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Responsible Party: Principal Investigator, Dr.A.Kranthi, PG Student, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: kranthirecession
Record Dates: First submitted 2018-08-20; First posted 2018-08-31 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Gingival Recession, Localized
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: The patients will be equally divided into two test groups. Group A and Group B after phase I therapy. the group A patients will be treated with laterally repositioned flap to obtain root coverage using microsurgical approach. The group B patients will be treated with laterally repositioned flap to obtain root coverage using macrosurgical approach
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Group A-15 patients were allocated to the microsurgical group for root coverage. following scaling and root planning, the laterally repositioned flap was done using the microsurgical approach
  Group B-15 Patients were allocated to the conventional group for root coverage following scaling and root planning, the laterally repositioned flap was done using the macrosurgical approach
  Interventions: Procedure: root coverage

INTERVENTIONS:
Procedure: root coverage — Group A: After administration of local anaesthesia using ophthalmic microsurgical knives a V-shaped incision was made in the gingival recession area. the gingiva was removed .the adjacent partial thickness pedicle flap was reflected from the donor area .the pedicle flap was then covered over the recipient site. then secured with 6-0 absorbable sling suture without tension. the surgical procedure was done with seilar microscope 40X magnification.
  Group B: After administration of local anaesthesia using 15 no blade a V-shaped incision was made in the gingival recession area . gingiva was removed .the adjacent partial thickness pedicle flap was reflected from the donor area .the pedicle flap was then covered over the recipient site. then carefully secured with 4-0 absorbable sling suture

SUMMARY:
This study was conducted to assess the evaluation of micro and Macro surgical approach in the treatment of grade II gingival recessions using the laterally repositioned flap

DETAILED DESCRIPTION:
In this study total, 30 patients were selected The patients initially received a comprehensive periodontal examination and complete plaque control program including oral hygiene to eliminate habits related to the aetiology of recession. Scaling, root planning and occlusal adjustments were done The patients were randomly assigned and divided into two groups. Group A and Group B. Patients with miller class II were treated with a laterally repositioned flap to obtain root coverage using conventional macrosurgical approach (15patients) and microsurgical approach(15patients)

The clinical parameters evaluated were height of gingival recession relative clinical attachment level which was measured as the distance from a fixed point in a stent to the bottom of the pocket and gingival biotype at baseline, 3 months and 6 months period

ELIGIBILITY:
Inclusion Criteria:

* Age 20-50 yrs
* ClassII gingival recession
* Vital teeth that were free from caries or inadequate restorations
* Sufficient width of attached gingiva

Exclusion Criteria:

* Any systemic diseases and smokers
* ClassI,III&IV gingival recession
* Abnormal frenal attachments
* Interdental bone loss with tooth mobility

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-08-16 (Actual)

PRIMARY OUTCOMES:
vertical depth of recession | Change in level of gingival margin from baseline to 6 months.
  The height of gingival recession: From cementoenamel junction to the free gingival margin.

SECONDARY OUTCOMES:
horizontal width of recession | Change in horizontal dimension of gingival margin from baseline to 6 months.
  The width of gingival recession: Horizontal dimension of gingival defect at the level of Cementoenamel junction..

CONTACTS AND LOCATIONS:
Overall Officials: veerendranath reddy, MDS, Study Director — panineeya mahavidyalaya institute of dental sciences
Locations (1):
- Panineeya Mahavidyalaya Institute of Dental Sciences, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Nizam N, Bengisu O, Sonmez S. Micro- and macrosurgical techniques in the coverage of gingival recession using connective tissue graft: 2 years follow-up. J Esthet Restor Dent. 2015 Mar-Apr;27(2):71-83. doi: 10.1111/jerd.12124. Epub 2014 Nov 13. PMID 25393983